CLINICAL TRIAL: NCT02998034
Title: Randomised Controlled Trial of Cemented Hemiarthroplasty Versus Uncemented Furlong Hemiarthroplasty
Brief Title: Cemented Hemiarthroplasty Versus Uncemented Furlong Hemiarthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peterborough and Stamford Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Martyn J Parker, Consultant orthopaedic surgeon, Peterborough and Stamford Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/WM/0049
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2018-04

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented monoblock hemiarthroplasty (Experimental): The cemented monoblock hemiarthroplasty is a double tapered polished stem with a hemiarthroplasty head cemented in place (Zimmer incorporated, UK)
  Interventions: Device: Cemented tapered stem hemiarthroplasty
- Hyroxyapatite coated prosthesis (Experimental): the Furlong Hyroxyapatite coated prosthesis (JRI orthopaedics limited UK) is a hydroxyapatite coating uncemented a hip prosthesis with a hemiarthroplasty head. The implant is uncemented.
  Interventions: Device: Uncemented Furlong Hemiarthroplasty

INTERVENTIONS:
Device: Uncemented Furlong Hemiarthroplasty — A furlong uncemeneted hyroxyapatite coated prosthesis.The hydroxyapatite stimulates bone ingrowth around the prosthesis and is this is thought to reduce loosening of the implant, residual pain and the long-term revision rate.
  Arms: Hyroxyapatite coated prosthesis
Device: Cemented tapered stem hemiarthroplasty — A cemented double tapered stem hemiarthroplasty
  Arms: Cemented monoblock hemiarthroplasty

SUMMARY:
In England each year over 9,000 people fracture their hip. Most of these are elderly females with the fracture occurring after a fall. Approximately half of these fractures are classified as intracapsular fractures because of their close proximity to the hip joint. The majority of these fractures are treated surgically by excising the broken femoral neck and removing the femoral head (ball part of the hip joint) and replacing it with an artificial hip joint. This hip replacement has traditionally been a hemiarthroplasty or sometimes termed a 'half hip replacement' in which only the ball part of the hip joint is replaced.

There are a number of different designs of hemiarthroplasty that may be used. Some of the implants are fixed in place with bone cement whilst the rest are inserted as a press fit without the bone cement. The early designs of implant were all press fit but these designs have now been shown to be inferior to those implants that are fixed in place with bone cement.

There are however a number of newer designs of implant that are coated with a substance (hydroxyapatite) that encourage the bone to grow onto the implant to fix it into place. To date these implants have only been compared to the cement fit implants in only one previous study. This study found no notable difference between the two types of hemiarthroplasty. This study aims to add to the research studies by comparing standard cement fit implant with a hydroxyapatite coated press fit implant to assist in determining the optimum surgical treatment for this common and disabling condition.

Both implants to be used in this study are still being used extensively within the United Kingdom and worldwide to treat this fracture. The study is therefore using two different implants within their recommended area of use, but in which there is uncertainty as to which is the best implant.

DETAILED DESCRIPTION:
As a follow-on from our current randomised trials of different types of treatment for hip fractures, we wish to undertake a prospective randomised trial to compare a modern cemented hemiarthroplasty prosthesis with a modern hydroxyapatite coated uncemented arthroplasty.

Cemented Exeter monoblock hemiarthroplasty The Exeter stemmed total hip replacement is considered one of foremost performing hip replacements in the world. The ETS (Exeter trauma stem) is one such implant and costs around £200. The implant has modern instrumentation and the stem has proven long term survival rates when used for total hip replacement.

Hyroxyapatite coated prosthesis Coating a hip prosthesis with hydroxyapatite is common practice for an uncemented hip replacement arthroplasty. The hydroxyapatite stimulates bone ingrowth around the prosthesis and is this is thought to reduce loosening of the implant, residual pain and the long-term revision rate.

The aim of the study is to assist in defining the optimum choice of arthroplasty for an acute hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Peterborough City Hospital with a displaced intracapsular fracture will be considered for inclusion in the study.

Exclusion Criteria:

* • Younger patients in which internal fixation is felt to be the choice of treatment to preserve the femoral head. This is generally those aged less than 60 years in which these patient have an expected good long term survival and are all treated by reduction and internal fixation.

  * All other patients in whom the injury is to be treated by reduction and internal fixation for a specific indication.
  * Those patients who are able to walk independently out of doors with no more than the use of a stick and are not cognitively impaired. These patients will first be considered for the ongoing randomised trial of Hemiarthroplasty or Total hip replacement (R&D reference - R&D/2012/30, REC reference - 12/LO/15490)
  * Patients who decline to participate.
  * Patients admitted when MJP is not available to supervise treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
regain of mobility | assessed at one year from injury
  measurement with a mobility score - Kristensen MT, Bandholm T, Foss NB, Ekdahl C, Kehlet H. High inter-tester reliability of the new mobility score in patients with hip fracture. J Rehabil Med 2008;40:589-91.

CONTACTS AND LOCATIONS:
Locations (1):
- Peterborough and Stamford Hospital NHS Foundation Trust, Peterborough, Cambs, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no IPD will be generated

REFERENCES:
- [Background] Parker MJ, Cawley S. Cemented or uncemented hemiarthroplasty for displaced intracapsular fractures of the hip: a randomized trial of 400 patients. Bone Joint J. 2020 Jan;102-B(1):11-16. doi: 10.1302/0301-620X.102B1.BJJ-2019-1041.R1. PMID 31888358